CLINICAL TRIAL: NCT00098215
Title: Pediatric Residency Training on Tobacco
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 1R01HD40683-1; 1R01HD040683 (NIH)
Record Dates: First submitted 2004-12-03; First posted 2004-12-06 (Estimated); Last update posted 2005-11-10 (Estimated); Status verified 2004-12

CONDITIONS: Tobacco Use Disorder
Keywords: Residency training
MeSH Terms: conditions — Tobacco Use Disorder

INTERVENTIONS:
Behavioral: Pediatric residency training on tobacco

SUMMARY:
The purpose of this study is to determine whether a specialized, technology-based training program in tobacco prevention is more effective than standard training for pediatric residents who counsel youth and their parents.

DETAILED DESCRIPTION:
The American Academy of Pediatrics and other leading health agencies call upon pediatricians to address environmental tobacco smoke (ETS), prevent smoking onset in youths, and encourage cessation of tobacco use by adolescents and their parents. Systematic intervention on tobacco by pediatricians would protect infants and young children from the harmful effects of ETS and save adolescents from a lifetime of addiction and tobacco-related disease. Despite this, few pediatricians address tobacco use, and pediatric residency training programs are not preparing residents to play a leadership role in the anti-tobacco arena.

The Pediatric Residency Training on Tobacco project is a four-year randomized controlled study of the efficacy of a specialized tobacco intervention program for pediatric residents. Eight participating pediatric training sites were randomly assigned to a Special Training condition featuring "Solutions for Smoking", a hybrid CD-ROM/Website training program. Six sites were randomly assigned to a control condition that provided standard print literature. Key features of "Solutions for Smoking" include a website containing background material on tobacco, interviewing, behavioral and pharmacological aspects of intervention, and a series of CD-ROMs containing audio-visual vignettes that model state-of-the-art interviewing and tobacco intervention skills. Residents are expected to practice the interventions with patients in their Continuity Clinics, and all sites are provided with brochures and other intervention materials for this purpose. Study investigators meet with residents at all sites three times per year to discuss the program and the residents' efforts to intervene on tobacco with their patients. Annually, second and third-year residents participate in Objective Structured Clinical Examinations (OSCEs) and a Resident Tobacco Survey. Patients and parents attending each of the Continuity Clinics complete Patient and Parent Tobacco Surveys at baseline and end of study.

Primary endpoints include changes over time in pediatric residents' tobacco intervention knowledge, skills, and activities as reported on the Tobacco Surveys and measured by performance on the OSCEs at baseline and follow-up. Secondary endpoints include changes in smoking, other tobacco use, and control of ETS by patients and parents. The study hypothesizes that pediatric residents in both arms of the study will be similar in knowledge and skills at baseline; that residents in the specialized training program will acquire more knowledge and greater skills for tobacco intervention during the course of the study compared to residents in the control condition; and residents in each condition will increase the frequency in which they address tobacco in patients and parents.

ELIGIBILITY:
The training program will include all residents enrolled in the 14 participating residency training programs.

The Baseline and Follow-up Resident Tobacco Surveys and OSCEs will include all second and third year residents enrolled in the residency training programs at baseline and years 1, 2, and 3 of follow-up.

The Baseline and Follow-up Patient Tobacco Survey will include 30 patients, ages 12-21, who were present in the waiting areas of the Continuity Clinic when the surveys were administered. All patients present in the clinic will be approached and invited to participate. Partcipants must be able to read English or Spanish, and patients who are attending the clinic for the very first time will not be eligible to participate in the survey.

The Baseline and Follow-up Parent Tobacco Surveys will be administered to 100 parents (one per family) who are present in the clinic when the surveys are administered. Parents who cannot read English or Spanish and who are bringing their child to the clinic for the very first time will not be able to participate.

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4000
Dates: Start 2001-03; Study Completion 2006-02

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Schwab, M.D., Principal Investigator — New Jersey Medical School
Locations (14):
- United States (14):
  - UMDNJ-Robert Wood Johnson Medical School, Camden, New Jersey
  - Mount Sinai School of Medicine (Jersey City Program), Jersey City, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Long Island College Hospital, Brooklyn, New York
  - Woodhull Medical and Mental Health Center, Brooklyn, New York
  - Brooklyn Hospital Center Program, Brooklyn, New York
  - Nassau County Medical Center, East Meadow, New York
  - New York Flushing Hospital Medical Center, Flushing, New York
  - Winthrop-University Hospital Program, Mineola, New York
  - New York and Presbyterian Hospital (Cornell Campus) Program, New York, New York
  - Lincoln Medical Center, The Bronx, New York
  - Bronx/Lebanon Hospital, The Bronx, New York